CLINICAL TRIAL: NCT06558708
Title: A Phase II Trial Comparing Efficacy, Tolerability, and Safety of GZR101 Injection and GZR33-70 Injection in Type 2 Diabetes Inadequately Controlled on Basal Insulin or Premixed Insulin Once Daily at Least With or Without Pre-dinner Meal-time Insulin
Brief Title: A Trial Comparing Efficacy, Tolerability, and Safety of GZR101 Injection Once Daily (OD) and GZR33-70 Injection OD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR101-T2D-202
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR101 Injection (Experimental): Participants will receive once daily GZR101 Injection with or without pre-dinner meal-time insulin, s.c, treat-to-target dose
  Interventions: Drug: GZR101 Injection
- GZR33-70 Injection (Experimental): Participants will receive once daily GZR33-70 Injection with or without pre-dinner meal-time insulin, s.c., treat-to-target dose
  Interventions: Drug: GZR33 Injection; Drug: Insulin aspart

INTERVENTIONS:
Drug: GZR101 Injection — Once daily
  Arms: GZR101 Injection
Drug: GZR33 Injection — Once daily
  Arms: GZR33-70 Injection
Drug: Insulin aspart — Once daily
  Arms: GZR33-70 Injection

SUMMARY:
This trial is conducted in China. The aim of the trial is to compare the efficacy, tolerability, and safety of GZR101 Injection and GZR33-70 Injection in type 2 diabetes inadequately controlled on basal/ premixed insulin once daily at least with or without pre-dinner meal-time insulin.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed the informed consent form (ICF) before the trial, fully understanding the trial content, process and possible adverse reactions, and being able to comply with the contraindications and restrictions specified in this protocol.
* 2.At the age of 18-75 (inclusive) at the time of informed consent, male or female.
* 3.Negative pregnancy test results for serum human chorionic gonadotropin (HCG) in women of childbearing potential at screening.
* 4.Diagnosed with type 2 diabetes mellitus above or equal to 6 months.

Exclusion Criteria:

* 1.Presence or history of malignant neoplasm prior to screening.
* 2.Known or suspected hypersensitivity to investigational medical product(s) or related products.
* 3.Severe hypoglycemia (Level 3 hypoglycemia) within 6 months prior to screening.
* 4.History of acute heart failure within 6 months prior to screening or hospitalization for coronary heart disease, myocardial infarction, unstable angina, stroke within 6 months prior to screening.
* 5. Participated in another interventional clinical study within 4 weeks prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0, week 16
  Change from baseline in HbA1c (Glycosylated Haemoglobin) after 16 weeks of treatment

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) | Week 0, Week 16
  Change from baseline in fasting plasma glucose (FPG) after 16 weeks of treatment
Change in 7-point SMPG profile | Week 0, Week 16
  Change from baseline in 7-point SMPG profile after 16 weeks of treatment: the mean and the CV
Incidence and Rate of Treatment-emergent AE/SAEs | Week 0, Week 19
  A TEAE is defined as an event that had onset date (or increase in severity) during the on-treatment observation period.
Incidence and Rate of hypoglycemia Events | Week 0, Week 19
  Hypoglycaemia alert episodes (level 1) are defined as episodes that are sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy with plasma glucose value of equal to or above (>=) 3.0 and less than (<) 3.9 mmol/L (>= 54 and < 70 mg/dL) confirmed by BG meter. Clinically significant hypoglycaemic episodes (level 2) are defined as episodes that are sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) are defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Severe hypoglycaemic episodes (level 3) are defined as episodes that are associated with severe cognitive impairment requiring external assistance for recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Study Site 01, Tianjin, China

IPD SHARING:
Plan to Share IPD: No